CLINICAL TRIAL: NCT01809522
Title: Does the Posterior Reconstruction of the Rhabdosphincter Improve Early Recovery of Continence After Robotic-Assisted Radical Prostatectomy? A Multicenter Randomized Controlled Trial. A Phase III Open-label Prospective International Multicenter Randomized Controlled Study for the Evaluation of the Efficacy of PRR, in Patients Subjected to RALP, Measured in Terms of Early Recovery of the Continence.
Brief Title: Does Posterior Reconstruction of the Rhabdosphincter Improve Early Recovery of Continence After Robotic-Assisted Radical Prostatectomy?
Acronym: PRR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Bernardo Rocco, Principal Investigator, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Posterior Reconstruction
Record Dates: First submitted 2013-03-09; First posted 2013-03-12 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Urinary Incontinence
Keywords: Robotic-assisted radical prostatectomy; Urinary continence; Posterior reconstruction of the rhabdosphincter; Posterior musculofascial plate reconstruction
MeSH Terms: conditions — Urinary Incontinence

ARMS (2):
- Posterior reconstruction of the musculofascial plate (Experimental): These patients will receive reconstruction of the muscolofascial plate after radical prostatectomy. The reconstruction will be performed using two 3-0 Poliglecaprone sutures (on RB-1 needles) tied together, with each individual length being 12-15 cm. seven - Ten knots will be placed when tying the sutures to provide a bolster. The free edge of the remaining Denonvillier's fascia will be identified after the prostatectomy and approximated to the posterior aspect of the rhabdosphincter and the posterior median raphe using one arm of the continuous suture. As a rule, four passes will be taken from the right to the left and the suture is locked. The second layer of the reconstruction will be then performed with the other arm of the suture approximating the posterior lip of the bladder neck (full thickness) and the vesicoprostatic muscle to the posterior urethral edge and to the already reconstructed median raphe .This suture will be then tied to the end of the first suture arm.
  Interventions: Procedure: Posterior reconstruction of the rhabdosphincter
- Standard radical prostectomy (No Intervention)

INTERVENTIONS:
Procedure: Posterior reconstruction of the rhabdosphincter
  Arms: Posterior reconstruction of the musculofascial plate

SUMMARY:
The present study is a multicenter randomized, controlled trial, whose aim is to verify the effect of the posterior reconstruction of the rhabdosphincter after robot-assisted radical prostatectomy on early recovery of urinary continence.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤ 80 years;
* Biopsy proven clinically localized prostate cancer;
* Informed consent obtained and signed;
* Understanding of, and willingness to comply with, the study procedures.

Exclusion Criteria:

* Pre-operative incontinence;
* Salvage prostatectomy (defined as a prostatectomy prescribed after the failure of a different primary treatment);
* Surgical posterior plane at the peri - rectal fat, without preserving an edge of the Denonvilliers;
* History of psychiatric or addictive disorder or other medical condition that, in the opinion of the investigator, would preclude the patient from meeting the trial requirements;

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Urinary continence | 12 months
  No urinary leakages, assessed with the EPIC Questionnaire.

SECONDARY OUTCOMES:
Oncologic radicality | 12 months
  PSA < 0,2 ng/ml.
Sexual potency | 12 months
  Potency sufficient for intercourse, with or without use of PDE5i, assessed with the IIEF Questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Milan, Italy